CLINICAL TRIAL: NCT05277623
Title: Effect of Mannitol on Postreperfusion Syndrome During Living Donor Liver Transplant: a Randomized Clinical Trial
Brief Title: Effect of Mannitol on Postreperfusion Syndrome During Living Donor Liver Transplant
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R 42/ 2022
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Liver Transplant Disorder
MeSH Terms: interventions — Mannitol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mannitol group (Active Comparator)
  Interventions: Drug: Mannitol
- control group (Placebo Comparator)
  Interventions: Other: 0.9% normal saline

INTERVENTIONS:
Drug: Mannitol — During the anhepatic phase, the patients in the mannitol group (30) will receive 1 g/kg
  Arms: mannitol group
Other: 0.9% normal saline — the same amount of 0.9% normal saline
  Arms: control group

SUMMARY:
Postreperfusion syndrome during living liver transplants remains a serious concern for transplant anesthesiologists. This syndrome is responsible for decreases in systemic blood pressure, systemic vascular resistance, and cardiac output and can even lead to cardiac arrest. Delayed graft function and primary graft nonfunction are closely related to postreperfusion syndrome (Therefore, attenuating the syndrome during anesthesia is of great importance.

ELIGIBILITY:
Inclusion Criteria:

* patients with end-stage liver disease who will undergo living donor transplantation.

Exclusion Criteria:

* Patients with a history of portopulmonary hypertension.
* Hepatopulmonary syndrome.
* Cirrhotic cardiomyopathy.
* Hepatorenal syndrome types 1 and 2.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
mean arterial blood pressure | one hour after reperfusion
  postreperfusion mean blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine Ain Shams University, Cairo, Egypt